CLINICAL TRIAL: NCT00889564
Title: HeRO Vascular Access Device Bacteremia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: Integra Clinical Trial Solutions - statistical analysis (Unknown); Ross, John, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-0050
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Hemodialysis
Keywords: Vascular access for hemodialysis; Catheter dependent patients; Access challenged patients; Bacteremia; HeRO Vascular Access Device
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: HeRO Vascular Access Device — Long-term subcutaneous vascular access device for hemodialysis

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of the HeRO Vascular Access Device in access challenged (e.g., catheter-dependent) hemodialysis patients. It is hypothesized the bacteremia rate associated with the HeRO device will be lower than a historical literature control of tunneled dialysis catheters.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older.
2. Male or non-pregnant female.
3. Life expectancy less than 1 year.
4. ESRD on hemodialysis with poor remaining venous access sites for creation of an AV fistula or placement of a graft in the upper extremities.
5. Implant side central venous system that surgeon believes can be accessed with interventional devices and can accommodate the 19 Fr GVAS device.
6. Potential GVAS target brachial artery ≥ 3 mm in diameter determined by any suitable measure.
7. Ability to understand and provide written informed consent.
8. Willing and able to cooperate with follow-up examinations.

Exclusion Criteria:

1. Documented history of drug abuse within six months prior to enrollment.
2. "Planned" concomitant surgical procedure or previous major surgery within 30 days, excluding vascular access related procedures.
3. Currently being treated with another investigational device or drug.
4. Known bleeding diathesis or hypercoaguable state.
5. Peripheral white blood cell count 1.5 K/mm3 or platelet count 50 K/mm3.
6. Degenerative connective tissue disease, e.g., Marfan's and Ehlers Danlos Syndrome. Subjects with Lupus Erythematosus may be enrolled if receiving no immunosuppressants or low dose prednisone only (< 10 mg/day orally).
7. Subjects with known or suspected concomitant active bacterial, fungal, viral, or parasitic infection. Subjects with Hepatitis B and/or Hepatitis C may be enrolled. Subjects who are HIV + with CD4 count of < 200 are excluded. Subjects with bacteremia within the past six (6) weeks must have negative blood cultures one week after completing appropriate antibiotic therapy prior to enrollment.
8. Severe underlying co-morbidity or immediate life-threatening condition.
9. Subjects with any condition which, in the opinion of the investigator, could preclude evaluation of response or completion of follow-up or affect subject safety.
10. Subjects with significant arterial occlusive disease which would preclude safe placement of an upper extremity hemodialysis access.
11. Subjects with history or findings on physical examination suggesting significant arterial insufficiency that could affect patient safety and/or device performance in the extremity planned for use with GVAS (i.e., steal syndrome, hand ischemia, peripheral arterial vascular disease, etc.).
12. Subjects with scheduled kidney transplant within the next 12 months.
13. Subjects with history of superior vena cava syndrome are excluded unless it was induced by previous access (these subjects can be enrolled).
14. Subjects with history of decreased cardiac output with ejection fraction < 20% and/or NYHA class III or IV. NYHA definitions: Class III - Subjects with marked limitation of activity; they are comfortable only at rest; Class IV - Subjects who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.
15. Subjects with history of uncorrected hypotension with systolic blood pressures routinely < 100 mg Hg.
16. Subjects who currently have a pacemaker or ICD in their central venous system on the same side where the GVAS device would be implanted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
HeRO superiority in device and implant procedure-related bacteremia compared to historical tunneled dialysis catheter literature control | 12 months

SECONDARY OUTCOMES:
Incidence of serious device or implant procedure-related serious adverse events and loss of secondary patency | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Ross, MD, Principal Investigator — Bamberg County Hospital
Locations (7):
- United States (7):
  - University of Miami / Cedars Medical Center, Miami, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - Southern Illinois University, Springfield, Illinois
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Bamberg County Hospital, Bamberg, South Carolina
  - Baptist Medical Center, San Antonio, Texas
  - Sentara Heart Hospital, Norfolk, Virginia